CLINICAL TRIAL: NCT03024775
Title: Clinical Response and Cytokines Production After Challenge With Different Wheat Genotypes in Patients With Not-celiac Wheat Sensitivity.
Brief Title: Response to Different Wheat Genotypes in Not-celiac Wheat Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ACPM16
Record Dates: First submitted 2016-12-30; First posted 2017-01-19 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac Wheat Sensitivity; ancient wheats; modern wheats; ATIs
MeSH Terms: interventions — Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (4):
- Active Comparator 1 (Active Comparator): Wheat flour with high inflammatory response will be administered blindly versus placebo for 15 days in NCWS patients.
  Interventions: Dietary Supplement: Wheat flour
- Active Comparator 2 (Active Comparator): Wheat flour with low inflammatory response will be administered blindly versus placebo for 15 days in NCWS patients.
  Interventions: Dietary Supplement: Wheat flour
- Placebo 1 (Placebo Comparator): Placebo (xylose) will be administered blindly versus wheat flour with high inflammatory response for 15 days in NCWS patients.
  Interventions: Dietary Supplement: Placebo
- Placebo 2 (Placebo Comparator): Placebo (xylose) will be administered blindly versus wheat flour with low inflammatory response for 15 days in NCWS patients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wheat flour — Wheat flour will be administered three times per day for 15 days.
  Arms: Active Comparator 1; Active Comparator 2
Dietary Supplement: Placebo — Placebo (xylose) will be administered three times per day for 15 days.
  Arms: Placebo 1; Placebo 2

SUMMARY:
Non-celiac gluten sensitivity (NCGS) is a condition where intestinal and extraintestinal symptoms are triggered by gluten ingestion in the absence of celiac disease and wheat allergy. Despite the great interest in NCGS, much remains unknown about the pathogenesis. Some studies seem to suggest that wheat components other than gluten (i.e. amylase/trypsine inhibitors, ATIs) can cause the symptoms, and therefore the term "non-celiac wheat sensitivity" (NCWS) has been proposed instead of NCGS. It is believed that this condition is worldwide increasing, due to the evolution of wheat breeding (i.e. consumption of wheats with high gluten content), and that ancient wheats are better tolerated by NCWS patients than the modern ones. Therefore, the aim of the study is to determine whether the common belief regarding the fact that ancient wheats are better tolerated by NCWS patients than the modern ones is confirmed by scientific data, and to identify the wheat kernel components triggering this pathology. The availability of wheat materials with opposite characteristics, such as the period of development (ancient vs. modern), or the technological properties (cultivars with weak glutens vs. strong gluten), or the presence/absence of specific ATIs polypeptides, will allow to define the role played by these factors. Therefore, the study has two objectives: 1) extraction and testing of total kernel proteins, in order to evaluate the inflammatory response to gluten and non-gluten proteins by peripheral blood mononuclear cells (PBMC) and immunocytes extracted by the rectal mucosa of NCWS patients and healthy control subjects, and 2) clinically testing two wheat genotypes, selected on the basis of the previous in vitro studies, showing the highest and the lowest in vitro inflammatory response, in order to verify their effect in triggering NCWS symptoms.

DETAILED DESCRIPTION:
Non-celiac gluten sensitivity (NCGS) is a condition where intestinal and extraintestinal symptoms are triggered by gluten ingestion in the absence of celiac disease and wheat allergy. Despite the great interest in NCGS, much remains unknown about the pathogenesis. Some studies seem to suggest that wheat components other than gluten (i.e. amylase/trypsine inhibitors, ATIs) can cause the symptoms, and therefore the term "non-celiac wheat sensitivity" (NCWS) has been proposed instead of NCGS. NCWS pathogenesis has been attributed to very different mechanisms: innate or adaptive immunity, incomplete digestion and/or absorption of fermentable oligosaccharides and disaccharides, monosaccharides and polyols, and, finally, psychological effect. In addition, it is believed that this condition is worldwide increasing, due to the evolution of wheat breeding (i.e. consumption of wheats with high gluten content), and that ancient wheats are better tolerated by NCWS patients than the modern ones. Therefore, the aim of the study is to determine whether the common belief regarding the fact that ancient wheats are better tolerated by NCWS patients than the modern ones is confirmed by scientific data, and to identify the wheat kernel components triggering this pathology. The availability of wheat materials with opposite characteristics, such as the period of development (ancient vs. modern), or the technological properties (cultivars with weak glutens vs. strong gluten), or the presence/absence of specific ATIs polypeptides, will allow to define the role played by these factors. The researchers take into consideration different tetraploid wheat genotypes derived from the Italian breeding activity carried out during the 20th century in comparison with landraces, primitive and old wheat cultivars previously cultivated and used mostly in Southern Italy for pasta and bread production, together with an experimental genetically modified (GM) wheat line expressing a lower amount of ATIs. For the purpose of the study, the collection has been subdivided into 5 groups, according to the breeding period. Wheat genotypes will be also evaluated for several parameters: protein content, gluten index, quantitative analysis of ATIs proteins by Mass Spectrometry, etc. The project has two objectives, related to the influence of wheat consumption on health: 1) extraction and testing of total kernel proteins, in order to evaluate the inflammatory response to gluten and non-gluten proteins by peripheral blood mononuclear cells (PBMC) and immunocytes extracted by the rectal mucosa of NCWS patients and healthy control subjects, and 2) clinically testing two wheat genotypes, selected on the basis of the previous in vitro studies, showing the highest and the lowest in vitro inflammatory response, in order to verify their effect in triggering NCWS symptoms.

ELIGIBILITY:
Inclusion Criteria:

All the patients will meet the recently proposed criteria:

* negative serum anti-tissue transglutaminase and antiendomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* absence of intestinal villous atrophy
* IgE-mediated immunoallergic tests negative to wheat (skin prick tests and/or serum specific IgE detection)
* follow-up duration >12 months after the initial diagnosis
* at least two outpatient visits during the follow-up period.

Adjunctive criteria adopted in our patients will be:

* resolution of the gastrointestinal symptoms on a standard elimination diet, without wheat, cow's milk, egg, tomato, chocolate, or other food(s) causing self-reported symptoms
* symptom reappearance on DBPC wheat challenge, performed as described previously. As in previous studies, DBPC cow's milk protein challenge and other "open" food challenges will be also performed.

Exclusion Criteria:

Exclusion criteria will be:

* age <18 years
* positive EmA in the culture medium of the duodenal biopsies, even if the villi to crypts ratio in the duodenal mucosa was normal
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other organic gastrointestinal diseases (i.e. careful exclusion of Crohn's disease)
* concomitant treatment with steroids and/or antihistamines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory response to wheat genotypes by PBMC of NCWS patients and healthy control subjects. | Through study completion, an average of 6 months
  Cytokines evaluation in response to gluten and non-gluten proteins from total kernel proteins of different wheat genotypes (i.e. ancient vs. modern vs. genetically modified) by PBMC of patients with a definitive diagnosis of NCWS, at the end of the diagnostic Double-Blind Placebo-Controlled (DBPC) wheat challenge, and of healthy control subjects.
Inflammatory response to wheat genotypes by rectal immunocytes of NCWS patients and healthy control subjects. | Through study completion, an average of 6 months
  Rectal immunocytes evaluation in response to gluten and non-gluten proteins from total kernel proteins of different wheat genotypes (i.e. ancient vs. modern vs. genetically modified) by immunocytes extracted by the rectal mucosa of patients with a definitive diagnosis of NCWS, at the end of the diagnostic Double-Blind Placebo-Controlled (DBPC) wheat challenge, and of healthy control subjects.

SECONDARY OUTCOMES:
Clinical response to wheat genotypes in NCWS patients | Change from baseline at 2 weeks
  Symptoms evaluation before and after a 2 weeks challenge with two wheat genotypes showing the highest and the lowest in vitro inflammatory response in diagnosed NCWS patients on gluten-free diet. During the challenge periods, the severity of symptoms will be recorded: the patients will complete a 100mm visual analog scale, which assesses the specific symptoms they report. The challenges will be considered positive if the same symptoms which had been initially present will reappear after their disappearance on elimination diet.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Background] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Background] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Background] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Background] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Background] Spits H, Cupedo T. Innate lymphoid cells: emerging insights in development, lineage relationships, and function. Annu Rev Immunol. 2012;30:647-75. doi: 10.1146/annurev-immunol-020711-075053. Epub 2012 Jan 6. PMID 22224763
- [Background] Spits H, Di Santo JP. The expanding family of innate lymphoid cells: regulators and effectors of immunity and tissue remodeling. Nat Immunol. 2011 Jan;12(1):21-7. doi: 10.1038/ni.1962. Epub 2010 Nov 28. PMID 21113163
- [Background] Veldhoen M, Withers DR. Immunology. Innate lymphoid cell relations. Science. 2010 Oct 29;330(6004):594-5. doi: 10.1126/science.1198298. No abstract available. PMID 21030634